CLINICAL TRIAL: NCT07180004
Title: Relationship Between Proximal and Distal Muscle Strength and Upper Extremity Functional Skills in Patients With Parkinson Disease (pwPD)
Brief Title: Upper Extremity Functional Skills in Patients With Parkinson Disease (pwPD)
Acronym: pwPD
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: Parkinson
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: PARKINSON DISEASE (Disorder); Upper Extremity; Muscle Strength Development; Functional Skills
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/study group: Individuals between the ages of 40 and 75 diagnosed with idiopathic Parkinson's disease (n=40)
- 2/control group: Healthy individuals between the ages of 40-75 (n=30)

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease, characterized pathologically by the progressive loss of dopaminergic neurons in the substantia nigra and clinically by the presence of motor symptoms such as bradykinesia, resting tremor, and/or rigidity.Patients with Parkinson's disease (pwPD) often exhibit poor manual dexterity and decreased strength. Fine motor deficits seen in PD include an inability to control cognitive power/force, poor manual dexterity, and motor dysfunction, which includes difficulties achieving the angles, speed, and coordination required for basic movements. Anatomical strength, as detailed in activities of daily living (ADL), is an important indicator of motor characteristics and vitality.Studies have shown a strong relationship between postural control and fine motor functions. For high-quality distal movement, better proximal stabilization is necessary. During upper extremity functions, the body's center of gravity must shift with arm movements, allowing adaptation to changing gravity. Good trunk control is essential in this dynamic process of maintaining balance. Studies examining this link between trunk control, balance, and hand functions are available in the literature. Among these studies conducted in diverse populations, studies involving PD are very few. Investigating parameters such as grip strength, upper extremity dexterity, and reaction time in PD will fill the gap in the literature. Meta-analysis studies have shown that muscle strength and strength in individuals with PD are lower than in healthy individuals. Furthermore, muscle strength in PD has been shown to be related to functional capacity and disease severity. In light of all this information, our study was designed to investigate the relationship between upper body muscle strength, particularly proximal and distal, and manual dexterity in PD. In this direction, the aim of this study is to determine the relationship between proximal and distal muscle strength and upper extremity functional abilities in PD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 40-75 years, diagnosed with idiopathic PD according to the UK Parkinson's Disease Association Brain Bank criteria by a specialist neurologist, with a Modified Hoehn & Yahr (m-HY) scale stage ≤4, and with a Mini Mental State Examination score of ≥22 for those with training and ≥18 for those without training, and with no known disease, volunteered to participate in the study.
* Individuals with no other known neurological and/or systemic disease
* Individuals without any upper extremity contractures

Exclusion Criteria:

* Individuals with diagnosed and/or treated psychiatric illnesses who are considered unable to complete the tests.
* Those taking neuroleptic medications or antidepressants.
* Individuals with orthopedic conditions that interfere with manual dexterity tests, such as severe dyskinesia, carpal tunnel syndrome, tendon injuries, or finger amputations; rheumatological conditions such as rheumatoid arthritis and osteoarthritis; and individuals with any neurological condition other than PD.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged between 40 and 75 years (n=40±5) who applied to the Neurology Clinic of the Faculty of Medicine of the University Hospital, diagnosed with Idiopathic Parkinson's disease by a neurologist, having stage ≤4 on the Modified Hoehn&Yahr (m-HY) scale, and having scores of ≥22 in the educated and ≥18 in the uneducated according to the Mini Mental State Examination, and healthy individuals of a similar age group (n=30±5)
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Muscle Strength Measurement | first day of assesment
  The isometric strength measurement will be performed using a digital muscle strength measurement device (KFORCE KINVENT) for the bilateral serratus anterior, upper trapezius, latissimus dorsi, deltoid, supraspinatus, teres minor, subscapularis, and biceps brachii muscles of the upper extremity.
Grip Strength Measurement | first day of assesment
  A Jamar hand dynamometer (Baseline®) and a PinchMeter (Baseline Mechanical Pinch Gauge with Case, Blue, 30 lb) will be used for grip strength measurement.The isometric strength measurement will be performed using a digital muscle strength measurement device (KFORCE KINVENT) for the bilateral serratus anterior, upper trapezius, latissimus dorsi, deltoid, supraspinatus, teres minor, subscapularis, and biceps brachii muscles of the upper extremity.
  Grip Strength Measurement: A Jamar hand dynamometer (Baseline®) and a PinchMeter (Baseline Mechanical Pinch Gauge with Case, Blue, 30 lb) will be used for grip strength measurement.
The 9-Hole Peg Test (DDPT) | first day of assesment
  The 9-Hole Peg Test (DDPT) is a validated test for PD that measures manual dexterity in seconds based on performance. The test material consists of nine standard-sized small rods and a nine-hole platform. The test will be administered with the patient in a seated position. The patient will be asked to place nine rods in the round compartment of the box as quickly as possible into the holes of the box, starting from the edge farthest from the compartment. Once completed, immediately remove them from the compartment, starting from the edge closest to the compartment. The test will begin with the dominant hand, and the time will be measured with a stopwatch. The time will begin when the hand touches the rods and will end when the last rod is placed in the box. The same procedure will be applied to the other hand. In this study, the arithmetic average of the test times, repeated twice, will be recorded separately for each hand.

SECONDARY OUTCOMES:
Demographic Form | first day of assesment
  (Medical history (disease duration and symptoms), demographic information (age, height, weight, education level), habits, medications, level of dependency in mobility in daily life, use of assistive devices)
Modified Hoehn & Yahr (m-HY) scale | first day of assesment
  PD disability will be assessed with the m-HY scale: stage 1.0 (unilateral involvement only); stage 1.5 (unilateral and axial involvement); stage 2.0 (bilateral involvement without balance impairment); stage 2.5 (mild bilateral disease with improvement in the pull test); stage 3.0 (mild to moderate bilateral disease; some postural impairment; physically independent); stage 4.0 (severe disability; still able to walk or stand unaided). Symptom severity in PD was graded using the Unified Parkinson's Disease Rating Scale (UPDRS): part I (mental dysfunction and mood); part II (activities of daily living); part III (motor component); part IV (treatment-related complications)
Unified Parkinson's Disease Rating Scale (UPDRS) | first day of assesment
  Symptom severity in PD is rated using the Unified Parkinson's Disease Rating Scale (UPDRS). Several items on this scale assess upper extremity and hand function. The Activities of Daily Living section assesses handwriting, cutting food, and grasping utensils. The Motor section assesses finger tapping, hand movements, and rapid alternating hand movements. These test items are scored from 0 to 4, with 4 representing maximum impairment and 0 representing normal movement ability. The UPDRS is comprised of subsections: Section I (mental dysfunction and mood); Section II (activities of daily living); Section III (motor); and Section IV (treatment-related complications).
Mini Mental State Examination (MMSE) | first day of assesment
  This test was developed by Folstein in 1975. Its Turkish validity and reliability study was conducted by Güngen et al. in 2002 (18). The Mini Mental State Examination (MMSE), which is quite suitable for screening cognitive function in the elderly and assesses cognitive functions in five separate areas (orientation, registration, attention and calculation, recall, and language), is frequently used. A score below 24 on the MMSE indicates dementia, 24-26 indicates mild cognitive impairment, and 26 or above indicates normal cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel tat, Associate Professor, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (2):
- Turkey (Türkiye) (2):
  - Kahramanmaraş Sütçü imam University, Kahramanmaraş, onikişubat
  - Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Onikişubat

IPD SHARING:
Plan to Share IPD: No